CLINICAL TRIAL: NCT02022137
Title: Evaluation of the Effect of a Cereal Bar With Added Agave Fructans or Lactitol or Lactose, in Patients With Minimal Hepatic Encephalopathy
Brief Title: Fructans, Lactitol and Lactose in Minimal Hepatic Encephalopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, Study Principal Investigator, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GAS-588-12/13-1
Record Dates: First submitted 2013-12-16; First posted 2013-12-27 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Liver Cirrhosis
Keywords: Minimal hepatic encephalopathy; Hepatic encephalopathy
MeSH Terms: conditions — Liver Cirrhosis; Hepatic Encephalopathy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Red cereal bar (Experimental): It includes the intervention of the red cereal bar for the designation of the group.
  Interventions: Dietary Supplement: Red cereal bar
- Green cereal bar (Placebo Comparator): It includes the intervention of the green cereal bar for the designation of the group.
  Interventions: Dietary Supplement: Green cereal bar
- White cereal bar (Active Comparator): It includes the intervention of the white cereal bar for the designation of the group.
  Interventions: Dietary Supplement: White cereal bar

INTERVENTIONS:
Dietary Supplement: Red cereal bar — Consumption of the cereal bar with agave fructans or lactitol or lactose added each bar with 10 grams of dietary fiber and 1.2 grams of protein by weight and 20 to 30 grams of fiber.
  Arms: Red cereal bar
Dietary Supplement: Green cereal bar — Consumption of the cereal bar with agave fructans or lactitol or lactose added each bar with 10 grams of dietary fiber and 1.2 grams of protein by weight and 20 to 30 grams of fiber.
  Arms: Green cereal bar
Dietary Supplement: White cereal bar — Consumption of the cereal bar with agave fructans or lactitol or lactose added each bar with 10 grams of dietary fiber and 1.2 grams of protein by weight and 20 to 30 grams of fiber.
  Arms: White cereal bar

SUMMARY:
As an alternative for the treatment of Minimal Hepatic Encephalopathy (MHE) Agave fructans have shown prebiotic effects, and have shown to improve function of the digestive system, control and induce glycemic effect satiety. Therefore the impact of the fermentation of such prebiotic in the gut may contribute to improving health and quality of life of patients with MHE.

DETAILED DESCRIPTION:
Hepatic encephalopathy (HE) is a potentially reversible neuropsychiatric syndrome characterized by changes in cognitive function, behavior and personality of patients with chronic liver disease or cirrhosis. Increased concentration of ammonia is the main precipitant of encephalopathy and brain astrocytes are the main affected cells in the neuropathology of this disease. The toxicity of ammonia together with the neutrophil dysfunction and oxidative stress and inflammation secondary to infection, result in a progressive decline in quality of life and an increased risk of accidents for patients with this disease.

About 28% of patients with liver cirrhosis develop encephalopathy during the course of the disease and within this percentage, 84% will develop MHE. Currently, chronic liver diseases are the third leading cause of death in Mexico. The high prevalence suggests that HE could become a public health problem, with the 2020 projected figures of 1.5 million people with cirrhosis, which represents approximately 400 000 to 500 000 people with probable encephalopathy.

The usual treatment of MHE is the use of antibiotics or pro and prebiotics, these enhances the performance and quality of life of patients who have the disease. The general consensus has been using lactulose or lactitol as the first treatment options for MHE consistent with data from previous studies. However, the rate of adherence to treatment with lactulose and lactitol is low, especially in patients with MHE with no symptoms and lack of specific information about their problems, to adhere to medications that can cause diarrhea and flatulence.

In the last eight years functional ingredients have been studied as alternatives to the treatment of patients with MHE. In 2004, Liu et al showed that 25% chicory inulin (prebiotic) and this combined with probiotics improve the psychometric function of MHE patients. In similar studies conducted in 2007 and 2009 in which they used a formulation with a symbiotic fructo-oligosaccharides based chicory inulin and B. longum, showed improvement in psychometric tests applied to patients. In 2008, Bajaj et al showed that patients who consumed a yogurt with probiotics, showed significant changes in the degree of MHE.

As an alternative for treating the MHE we found Agave tequilana Weber fructans, which present prebiotic effect, besides having shown to improve the function of the digestive system, control and induce glycemic effect satiety. Therefore the impact of the fermentation of such prebiotic in the gut may contribute to improving the health and quality of life of patients with MHE.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 70 years.
* Liver cirrhosis of any etiology.
* Presence of minimal hepatic encephalopathy.
* Presence of hepatic encephalopathy I

Exclusion Criteria:

* Hepatic encephalopathy II or III
* Use of antibiotics in the previous month.
* Presence of immunological diseases.
* Consumption of probiotics.
* Patients with hepato-renal diseases.
* Patients who do not agree to participate in the project.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Minimal hepatic encephalopathy | 2 months
  Assessed by psychometric Hepatic Encephalopathy (PHES) and Critical Flicker Frequency (CFF)

SECONDARY OUTCOMES:
Nutritional Status | 2 months
  Measured with the following parameters:body weight and height (to calculate BMI), triceps skinfold and mid-arm circumference (to calculate mid-arm muscle circumference, and bioelectrical impedance vector analysis.

OTHER OUTCOMES:
Ammonia, liver function tests | baseline and 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Aldo Torre Delgadillo, M.D. M.Sc, Principal Investigator — INCMNSZ
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, México, D.f., Mexico